CLINICAL TRIAL: NCT00857207
Title: Metacognitive Training to Enhance Strategy Use in Blast Related TBI
Brief Title: Metacognitive Training to Enhance Strategy Use in Blast-Related TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0902-W
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Brain Concussion; Blast Injuries
Keywords: Cognitive Therapy; Outcomes Assessment
MeSH Terms: conditions — Brain Concussion; Blast Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Treatment Goal Management Training (Experimental): Treatment Goal Management Training
  Interventions: Behavioral: Goal Management Training
- Arm 2: Control-Brain Health Workshop (No Intervention): Control-Brain Health Workshop

INTERVENTIONS:
Behavioral: Goal Management Training — Enhanced Goal Management Training is a 10-week group therapy that teaches strategies to improve an individual's ability to complete everyday tasks.
  Arms: Arm 1: Treatment Goal Management Training

SUMMARY:
Enhanced Goal Management Training (GMT) is a 10-week group or individual therapy that teaches strategies to improve an individual's ability to complete everyday tasks. This research study will test the effect of GMT on 36 OEF/OIF Veterans compared to a control group of 16 OEF/OIF Veterans receiving a Brain Health Workshop. The results will provide information to conduct future research with a larger group of patients or to identify which patients demonstrate more benefit from the training.

DETAILED DESCRIPTION:
OBJECTIVES:

Aim 1: is to test benefits of GMT for improving executive function. Aim 2: Investigate factors which affect response to treatment.

RESEARCH PLAN:

This is a randomized controlled study to investigate the effect of Goal Management Training (GMT) for those with blast-related mTBI. The control group will participate in the Brain Health Workshop (BHW; Levine 2011), developed specifically for consistency with GMT session length and contact with the facilitator (Levine, 2011). Study outcome measures will be collected at pre- and post-treatment, and at 1 month after the end of treatment.

Family Member/Friend of Participant. The participant will identify a friend or family member who observes his/her everyday behavior at least 2-3 hours, twice a week. After obtaining the consent of the person, both the participant and his/her friend or family member(s) will attend a general education session about brain function and treatments. In addition to attending the education session the consenting friend or family member will answer a questionnaire (BRIEF-A) about the participant's executive function. The friend or family member will also receive phone calls weekly in order to report the participant's ease or difficulties in completing homework.

METHODS:

The investigators will enroll 54 participants, recruited from the North Florida/South Georgia Veteran Health System in Gainesville. Clinical staff will inform outpatients about the study. Patients interested in hearing more about the research study will be provided with contact information for the study staff. A meeting will be scheduled and candidates will be screened.

Participants will be randomly assigned to either treatment or control groups, in a ratio of 38:16. In addition, the Pocock-Simon covariate adaptive randomization procedure will be used so that, for each PTSD severity category within each of the two sites, approximately 70% (38/54) of subjects are assigned to treatment group; consequently, there will be approximately equal proportion of PTSD subjects assigned to the treatment and control groups within each of the two study sites.

Simulated Practice In The Laboratory: Training tasks include exercises such as: 1) clapping to words and inhibiting clapping to a targeted word; 2) card sorting; 3) decision making and planning in order to complete five activities within a four minute time span; 4) Catalog Task; and 5) Book keeping task. Initially, the exercises are relatively easy and subsequently progress to greater complexity. Participant's strengths and weaknesses are discussed. Improvements are identified and reinforced as they learn more efficient planning and problem solving. The following steps are taught during simulated tasks: 1) Identify Main Goal; 2) Break down task into sub-goals and steps for each goal; 3) List supplies needed; 4) Recognize potential barriers to completing goal; 5) Determine strategy to accomplish task: 6) Prepare to begin task with "presence of mind" exercise; 7) State goal out loud; 8) Begin task and stop self frequently to state main goal out loud and check to be sure one is working toward the goal (on target).

Functional Practice at Home and with Smartphone Technology: In addition to lab practice, the original GMT (Levine, 2000)includes three tasks that must be practiced at home. Participants identify a complex task with which they are having difficulty, for example, meal planning and shopping; planning a party; building a birdhouse; or paying monthly bills. Generalization of laboratory practice to home environment is of critical importance. Unfortunately, the original GMT did not provide a method to monitor the frequency or success of home practice, nor a method to support productive practice in the home environment. In prior work, the investigators developed The Veteran's Task Manager (A Smartphone application (AP). Participants will use the AP features to break down tasks, estimate time to complete, check off each step as completed, respond to the visual/vibrating alert of "Goal" and respond to alert if "On Target". Information will be collected by the AP, such as accuracy of planned steps, time to complete task, and number of distractions from goal. The AP will record the participant's performance in functional practice at home and this information will be reviewed at the next lab session.

Control Group Intervention. The Brain Health Workshop (BHW; Levine 2011) was developed specifically for consistency with GMT session length and contact with the facilitator (Levine, 2011). BHW is an education presentation on brain function and cognitive principles of learning. Information about stress reduction, sleep hygiene, energy management, exercise and communication are covered with homework and quizzes on information covered.

FINDINGS: Initial report

ELIGIBILITY:
Inclusion Criteria:

* 2 incidences of blast-related mTBI according to the American Congress of Rehabilitation Medicine, any of three following criteria:

  * loss of consciousness <30 minutes, a Glasgow Coma Scale of 13
  * loss of memory for events immediately before and after the event (24 hours alteration of mental state at the time of accident)
  * focal neurological deficits that may, or may not, be transient (ACRM, 1993)
* Diagnosis must be documented in the medical record by a physician or neuropsychologist.
* Frontal Lobe impairment will be determined by 1.5 standard deviations below the mean on either the D-KEFS Color Word Interference Testorthe EXAMINER composite score.
* Age 18 to 55 years.
* At least 6 months post injury.
* Family member or friend that is willing to answer questionnaires and provide feedback on questionnaires and completion of homework.

Exclusion Criteria:

* History of pre-morbid learning disability.
* History of psychiatric diagnosis sufficiently severe to have resulted in inpatient hospitalization.
* Neurological disease unrelated to TBI (seizure disorder, stroke, ADHD).
* Score < 90 on National Adult Reading Test.
* Failure of validity testing on the Test of Memory Malingering (TOMM)
* Reported alcohol or substance abuse within the past year, or such abuse documented in medical record.
* Reported involvement in current litigation.
* Changes within the past month of medications known to affect cognitive functions e.g. benzodiazepines, opioids, antidepressants and antipsychotics.
* Currently enrolled in other cognitive therapy that cannot be discontinued.
* Not fluent in English.
* Not competent to provide consent (also, not able to demonstrate understanding of expectations of study and potential risks of participation).
* Patients who receive > 5 hours of therapy from a mental health specialist during the study will not be included in the final analysis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia K. Waid-Ebbs, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Waid-Ebbs JK; BCBA-D; Daly J, Wu SS, Berg WK, Bauer RM, Perlstein WM, Crosson B. Response to goal management training in veterans with blast-related mild traumatic brain injury. J Rehabil Res Dev. 2014;51(10):1555-66. doi: 10.1682/JRRD.2013.12.0266. PMID 25860148

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: Control-Brain Health Workshop: Control-Brain Health Workshop
  Brain Health Workshop is a 10-week therapy that teaches information about how the brain works with equal contact to the therapist as Goal Management Training
Period: Overall Study
Arm/Group | Arm 1: Treatment Goal Management Training | Arm 2: Control-Brain Health Workshop
Started | 48 | 3
Completed | 14 | 3
Not Completed | 34 | 0
Not completed — Withdrawal by Subject | 13 | 0
Not completed — did not meet inclusion criteria for deficit in inhibition or failed the TOMM | 18 | 0
Not completed — Subject chose not to participate after signing consent | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Treatment Goal Management Training | Arm 2: Control-Brain Health Workshop | Total
Number analyzed (Participants) | 14 | 3 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (7.2) | 41.7 (4.2) | 38.98 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 12 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 0 | 4
  White | 9 | 2 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 3 | 17
Post-traumatic stress disorder checklist-military version [Mean (Standard Deviation); unit: units on a scale] — scores range from 0-85 with higher scores indicating worse outcome, or more problems with Post Traumatic Stress Disorder symptoms.
  units on a scale | 60.9 (16.4) | 64.3 (4.7) | 62.6 (14.86)
Beck's Depression Inventory-II [Mean (Standard Deviation); unit: units on a scale] — scores range from 0-63 with higher scores indicating worse outcome or more depressive symptoms
  units on a scale | 31 (12.2) | 25.7 (12.0) | 30.06 (11.97)
North American Reading Test Estimated Intelligence Quotion [Mean (Standard Deviation); unit: units on a scale] — NART estimated IQ ranges from 80.22 to 127.8 with higher scores indicating better IQ.
  units on a scale | 111.1 (7.02) | 104.4 (8.1) | 109.95 (7.22)

OUTCOME MEASURES:

1. Primary Outcome: Computerized Tower Of London (cTOL)
Description: a computerized program in which patients are shown two pictures simultaneously of a goal board and a test board and are instructed to use the fewest possible moves to match the two boards within 60 seconds. Each baseline and 10 week set of 30 problems consists of the same number of 4, 5, 6 or 7 move problems and has the same average difficulty level. The dependent variables are the total time spent solving the problem (0-60 seconds for each problem; less time is better) and the proportion of optimal moves (toward the goal 0-1 with 1 being the best outcome) and time to first move (0-60 seconds with more planning time indicating better outcome).
Time Frame: Baseline, 10 weeks
Population: t-test
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Arm 1: Treatment Goal Management Training | Arm 2: Control-Brain Health Workshop
Number analyzed (Participants) | 14 | 3
Seconds
  cTOL Total time baseline | 24.6 (5.37) | 25.1 (4.43)
  cTOL Total time post treatment | 21.7 (4.3) | 24.7 (1.68)
  cTOL Time to first move baseline | 7.98 (2.44) | 9.11 (0.79)
  cTOL Time to first move Post | 8.21 (2.01) | 12.6 (2.41)
Statistical Analysis 1: Comparison: Arm 1: Treatment Goal Management Training vs Arm 2: Control-Brain Health Workshop; Linear regression of change of cTOL time to first move in GMT versus BHW group; Test type: Superiority; p = 0.0004, Regression, Linear; dependent variable: post-treatment outcome; independent variables:pre-treatment measurement and group indicator; Mean Difference (Final Values) = -3.95, Standard Error of Mean 1.14
Statistical Analysis 2: Comparison: Arm 1: Treatment Goal Management Training; total time will significantly improve 10 weeks from post; Test type: Superiority; p = 0.012, t-test, 2 sided; Mean Difference (Final Values) = -2.92, Standard Deviation 3.55
Statistical Analysis 3: Comparison: Arm 1: Treatment Goal Management Training; Time to first move will significantly increase at 10 weeks from baseline to indicate better planning; Test type: Superiority; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = 0.02, Standard Deviation 2.04

2. Secondary Outcome: BRIEF-A
Description: Behavior Rating Inventory of Executive Functions-Adult (BRIEF-A) is a self and informant report questionnaire consisting of 75 statements about executive behaviors. There are three possible responses to items: often, sometimes, never. Two subscale scores behavioral regulation index and metacognitive index are reported as T-scores adjusted for age with a possible score of 0-100. Lower scores are better indicating less trouble with executive function.
Time Frame: Baseline, 10 weeks
Population: T-test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Treatment Goal Management Training | Arm 2: Control-Brain Health Workshop
Number analyzed (Participants) | 14 | 3
score on a scale
  BRIEF Metacognitive Index Baseline | 78.6 (11.1) | 70.3 (9.29)
  BRIEF-A Metacognitive Index Post | 75.9 (11.0) | 68.7 (20.5)
  BRIEF-A Behavioral Regulation Index Baseline BRIEF-A Behavioral Regulation Index Baseline | 72.1 (13.1) | 66.3 (3.79)
  BRIEF-A Behavioral Regulation Index Post | 69.5 (12.8) | 60.0 (13.5)
Statistical Analysis 1: Comparison: Arm 1: Treatment Goal Management Training; paired T-test, Behavioral Regulation Index will improve at week 10 from baseline; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = 2.64, Standard Deviation 6.42
Statistical Analysis 2: Comparison: Arm 1: Treatment Goal Management Training; paired t-test of Metacognitive Index, MI will improve at 10 weeks compared to baseline; Test type: Superiority; p = 0.24, t-test, 2 sided; Mean Difference (Final Values) = 2.79, Standard Deviation 8.4

3. Secondary Outcome: cTOL Optimal Moves
Description: computerized program in which patients are shown two pictures simultaneously of a goal board and a test board and are instructed to use the fewest possible moves to match the two boards within 60 seconds. Each baseline and 10 week set of 30 problems consists of the same number of 4, 5, 6 or 7 move problems and has the same average difficulty level. Optimal moves are a proportion of optimal moves (toward the goal 0-1 with 1 being the best outcome).
Time Frame: baseline, 10 weeks
Population: Veterans with mTBI
Measure: Mean (Standard Deviation); unit: proportion of optimal moves
Arm/Group | Arm 1: Treatment Goal Management Training | Arm 2: Control-Brain Health Workshop
Number analyzed (Participants) | 14 | 3
proportion of optimal moves
  Baseline Optimal Moves | 0.67 (0.13) | 0.71 (0.03)
  10 week Optimal moves | 0.71 (0.12) | 0.80 (0.07)
Statistical Analysis 1: Comparison: Arm 1: Treatment Goal Management Training; optimal moves will significantly increase at 10 weeks from baseline; Test type: Superiority; p = 0.30, t-test, 2 sided; Median Difference (Final Values) = 0.03, Standard Deviation 0.09

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Arm 1: Treatment Goal Management Training | Arm 2: Control-Brain Health Workshop
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/3
Other Adverse Events (participants affected / at risk) | 0/14 | 0/3

LIMITATIONS AND CAVEATS:
recruitment of the anticipated number of participants per arm was not reached due to the unexpected closure of one of the recruitment sites. The data analysis was conducted by combining participants from two pilot studies and the randomized study to increase the number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT00857207/Prot_SAP_000.pdf